CLINICAL TRIAL: NCT01315366
Title: Phase III Study on the Effect of Vitamin D Supplementation on Indices of Mineral and Musculoskeletal Metabolism and on Parameters of Glucose and Fuel Metabolism in Elderly Subjects
Brief Title: Hypovitaminosis D : A Link Between Bone/Mineral and Fat/Fuel Metabolism
Acronym: GEHF-VitD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: Hotel Dieu de France Hospital (Other); Rafic Hariri University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Ghada El-Hajj Fuleihan, Professor, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AUBMC-GE-HF-1; AUBMC-IM-GE-HF-20 (Other Grant/Funding Number: American University of Beirut)
Record Dates: First submitted 2011-02-02; First posted 2011-03-15 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-03

CONDITIONS: Hypovitaminosis D; Insulin Resistance; Obesity; Osteoporosis
Keywords: Vitamin D; Elderly; Cardiovascular profile; Insulin resistance; Gene polymorphisms
MeSH Terms: conditions — Vitamin D Deficiency; Insulin Resistance; Obesity; Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose vitamin D (Active Comparator): Ci-Cal D (1000mg/day) and vitamin D (500IU/day) Ci-Cal D daily, plus a supplement of vitamin D3 EuroD (20,000 IU/wk) for one year.
  Interventions: Dietary Supplement: Euro D and Ci-CalD
- Low dose Vitamin D (Placebo Comparator): Ci-Cal D (1000mg/day) and vitamin D (500IU/day) Ci-Cal D daily, plus a weekly placebo (EURO D Placebo) supplement for one year.
  Interventions: Dietary Supplement: Euro D, Ci-CalD

INTERVENTIONS:
Dietary Supplement: Euro D and Ci-CalD — Ci-Cal D (1000mg/day) and vitamin D (500IU/day) daily, plus a supplement of vitamin D3 (20,000 IU/wk) for one year.
  Other Names: Europharm
  Arms: High dose vitamin D
Dietary Supplement: Euro D, Ci-CalD — Ci-Cal D(1000mg/day) and vitamin D (500IU/day) Ci-CalD daily, plus a weekly placebo Euro D supplement for one year.
  Other Names: EuroPharm
  Arms: Low dose Vitamin D

SUMMARY:
The optimal dose of vitamin D needed to optimize beneficial effects on musculoskeletal outcomes remains to be defined. Equally unclear is the impact of vitamin D on fuel metabolism and insulin sensitivity in human subjects. Thus, the overall objective of this proposal is to test the hypothesis that in ambulatory overweight elderly individuals, vitamin D administration at doses higher than currently recommended will:

1. Have a salutary effect on parameters of glucose and fuel metabolism. It will thus decrease indices of insulin resistance, improve lipid profile, and decrease markers of cardiovascular disease including adipokines, inflammatory cytokines, and markers of cell adhesion.
2. Have a superior effect on indices of mineral and musculoskeletal metabolism, including bone remodeling markers, lean mass, and bone mineral density.

We will investigate whether this effect is modulated by entry status of vitaminD and PTH as detailed below

DETAILED DESCRIPTION:
It has become increasingly recognized that low vitamin D levels are prevalent worldwide and to a more severe degree in the Middle East. Low vitamin D levels are associated with an increased risk of osteoporotic fractures, and of chronic conditions such as autoimmune disorders, diabetes, cancer, and the metabolic syndrome. Obese individuals are more likely to have low vitamin D levels, and in some studies obesity was a risk factor for fractures in both the young and elderly. Our group has investigated the impact of vitamin D therapy in the young, and preliminary data suggest that doses exceeding the currently updated recommended estimated average requirement (EAR) of 400IU for that age group may be more beneficial for bone health. The updated EAR recommendations by the IOM for any age group, although believed to cover the needs of all individuals in each age group, are limited by the lack of good evidence supporting such recommendations. Therefore, to-date, the optimal dose of vitamin D for both the young and elderly is unknown.

Two hundred and fifty elderly (age≥65 years), overweight (BMI ≥25kg/m2) non-diabetic individuals, will be recruited through outpatient clinics that investigators may have access to at American University of Beirut-Medical Center (AUB-MC), Hotel Dieu de France (HDF) and Rafic Hariri University Hospital (RHUH), and will be randomized after a pre-screen, in a double-blinded fashion, to receive 500 IU or the equivalent of 3357 IU of vitamin D3 daily for one year. Clinical information, exercise questionnaires will be obtained at 0 and 12 months.In addition, subjects partaking in the original study will be offered the option to participate in the validity and reliability study of a food frequency questionnaire to assess dietary intakes of Ca, vitamins D and K, and to participate in the vascular study evaluating the relation of the above nutrients with vascular parameters. Information on educational level, insurance status, dietary, sunscreen use, sun exposure and skin pigmentation will be obtained at baseline. Information on falls, trauma, history of fractures and medications will be obtained at each visit (0, 3, 6 and 12 months). The measurement of height, weight, BMI, waist, hip, waist/hip ratio, mid arm circumference, mid-calf circumference and muscle strength of the subject, enrolled in the study, will be triplicated on each visit at 0,3,6 and 12 months. Blood pressure and heart rate will be measured at screening, baseline, 3 months, 6 months and 12 months. Blood will be drawn at baseline, 3, 6 and 12 months for measurement of serum creatinine, calcium, phosphorous, alkaline phosphatase, 25-OHD, 1,25(OH)2D, PTH, indices of bone remodeling (osteocalcin and crosslaps), and a second morning void urine specimen will be collected for Ca/Cr. Insulin resistance will be measured using the McAuley as well as HOMA and QUCKI indices. We will also measure serum levels of adipokines (adiponectin, leptin), DLK1-Pref1, inflammatory markers (CRP, IL-6) and adhesion molecules (sICAM, sVCAM). We will characterize polymorphisms of genes affecting mineral metabolism such as VDR, CaSR,ER and CYP2R1, and will measure adiponectin R expression from subcutaneous fat and muscle biopsies that will be obtained at 0 and 12 months.Bone density scans of Lumbar Spine, Femoral Neck, Total Hip, Total Body, Sub Total Body, body composition and hip structural analyses parameters as well as TBS variables for the spine will be obtained at the baseline and at 12 months of the study. A visit at 9 months will be scheduled to supply subjects with Ci-cal D and Euro D, and to ensure compliance. IRB approval and consent forms will be obtained. An independent Data and Safety Monitoring Board will be asked to review serious adverse events and if needed may be asked to review unblinded data at recruitment of 30%, 60% and 100% of study subjects and of serious adverse events forms throughout the study duration.Repeated measures analyses will be used to evaluate differences in outcomes of interest between the two treatment groups and time effect within each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Elderly subjects (> or equal to 65 years old)without any disease mentioned in the exclusion criteria.
* BMI ≥ 25Kg/meters squared

Exclusion Criteria:

* Exclusion criteria include: diabetes, subjects with impaired glucose tolerance on medication, presence of a chronic disease or major organ failure such as severe heart failure, kidney or liver failure, conditions or intake of medications known to affect bone metabolism, rickets or osteomalacia, history of kidney stones, a baseline vitamin D level of less than 10 ng/ml and history of fragility fractures or an overall fracture risk based on FRAX of >10% .
* Subjects with impaired glucose tolerance on no medications will not be excluded.
* The classification of individuals as diabetics or having impaired glucose tolerance will be based on the American Diabetes Association criteria for diagnosis.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 257 (Actual)
Dates: Start 2011-01; Primary Completion 2014-08 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The HOMA index of insulin resistance | 1 year
  A full assessment of insulin resistance will be performed,using the HOMA, McAuley and QUICKI indices.
  The impact of vitamin D on all outcomes of interest will be assessed by treatment arms and then in sub-group analyses:
  * by baseline levels of vit D-PTH at study entry: Vitamin D< 20 ng/ml-PTH>76pg/ml; vitamin D<20ng/ml and PTH<76 pg/ml, vitamin D>20ng
  * by gender
Bone mineral density (BMD) at the spine,hip and total body measured by DXA and bone turnover markers (Osteocalcin and cross laps). | 1 year
  We will measure the bone mineral density at the spine, hip and total body. We will also test the bone turnover markers as osteocalcin and cross laps.

SECONDARY OUTCOMES:
Insulin, C- peptide, Fasting glucose, Chemistries, Vitamin D metabolites, Vitamin D binding protein, Urinary Ca/Cr ratio ,serum lipids,inflammatory markers(IL-6, CRP),adhesion molecules (sVCAM), GLA-OC and GLU-OC. | 1 year
  Gamma-Carboxyglutamatic Osteocalcin (GLA-OC) and Undercarboxylated Osteocalcin (GLU-OC).
Body fat mass and body lean mass measured by DXA | 1 year
Serum DLk1 levels | 1 year
  Serum DLK1 levels Preadipocyte factor 1 (Pref-1), also known as delta like protein (Dlk1), is a molecule that belongs to the Notch Delta family of signaling molecules, epidermal growth factor (EGF)-like super family, and possesses several isoforms, some circulating, also termed Fetal antigen 1 (FA1).
Adiponectin Receptor expression and Leptin from subcutaneous fat and muscle biopsies at baseline and follow-up. | 1 year
Morphologic bone assessment gathered defined by techniques incorporated into BMD acquisition scan image: Hip structural analyses parameters (Cortical thickness, Cross-sectional moment of inertia, section modulus) and trabecular bone structure (TBS) | 1 year
Mc Auley Index of insulin resistance by subgroups of patients divided by polymorphisms of genes affecting mineral metabolism (VDR, ER, CaSR, and CYP2R1 gene polymorphisms). | 1 year
BMD at the hip and body composition by subgroups of patients divided by polymorphisms of genes affecting mineral metabolism (VDR, ER, CaSR, and CYP2R1 gene polymorphisms). | 1 year
Bone turnover markers by subgroups of patients divided by polymorphisms of genes affecting mineral metabolism (VDR, ER, CaSR, and CYP2R1 gene polymorphisms). | 1 year
Bone mineral density (BMD) at the spine measured by DXA | 1 year
Adiponectin Receptor expression from subcutaneous fat and muscle biopsies | 1 year
Morphologic bone assessment gathered defined by techniques incorporated into BMD acquisition image:Hip structural analyses parameters and trabecular bone structure by subgroups of subjects divided by polymorphisms of genes affecting mineral metabolism | 1 year
  Genes affecting mineral metabolism are VDR, ER, CaSR, and CYP2R1 gene polymorphisms

CONTACTS AND LOCATIONS:
Overall Officials: Ghada El Hajj Fuleihan, MD, MPH, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon

REFERENCES:
- [Background] Fuleihan GE, Deeb M. Hypovitaminosis D in a sunny country. N Engl J Med. 1999 Jun 10;340(23):1840-1. doi: 10.1056/NEJM199906103402316. No abstract available. PMID 10366324
- [Background] El-Hajj Fuleihan G, Nabulsi M, Tamim H, Maalouf J, Salamoun M, Khalife H, Choucair M, Arabi A, Vieth R. Effect of vitamin D replacement on musculoskeletal parameters in school children: a randomized controlled trial. J Clin Endocrinol Metab. 2006 Feb;91(2):405-12. doi: 10.1210/jc.2005-1436. Epub 2005 Nov 8. PMID 16278262
- [Background] Arabi A, Zahed L, Mahfoud Z, El-Onsi L, Nabulsi M, Maalouf J, Fuleihan Gel-H. Vitamin D receptor gene polymorphisms modulate the skeletal response to vitamin D supplementation in healthy girls. Bone. 2009 Dec;45(6):1091-7. doi: 10.1016/j.bone.2009.07.074. Epub 2009 Jul 30. PMID 19647104
- [Background] Lips P, Hosking D, Lippuner K, Norquist JM, Wehren L, Maalouf G, Ragi-Eis S, Chandler J. The prevalence of vitamin D inadequacy amongst women with osteoporosis: an international epidemiological investigation. J Intern Med. 2006 Sep;260(3):245-54. doi: 10.1111/j.1365-2796.2006.01685.x. PMID 16918822
- [Background] Arabi A, Baddoura R, Awada H, Salamoun M, Ayoub G, El-Hajj Fuleihan G. Hypovitaminosis D osteopathy: is it mediated through PTH, lean mass, or is it a direct effect? Bone. 2006 Aug;39(2):268-75. doi: 10.1016/j.bone.2006.01.140. Epub 2006 Feb 21. PMID 16495164
- [Background] Dobnig H, Pilz S, Scharnagl H, Renner W, Seelhorst U, Wellnitz B, Kinkeldei J, Boehm BO, Weihrauch G, Maerz W. Independent association of low serum 25-hydroxyvitamin d and 1,25-dihydroxyvitamin d levels with all-cause and cardiovascular mortality. Arch Intern Med. 2008 Jun 23;168(12):1340-9. doi: 10.1001/archinte.168.12.1340. PMID 18574092
- [Background] Parikh SJ, Edelman M, Uwaifo GI, Freedman RJ, Semega-Janneh M, Reynolds J, Yanovski JA. The relationship between obesity and serum 1,25-dihydroxy vitamin D concentrations in healthy adults. J Clin Endocrinol Metab. 2004 Mar;89(3):1196-9. doi: 10.1210/jc.2003-031398. PMID 15001609
- [Background] Pittas AG, Lau J, Hu FB, Dawson-Hughes B. The role of vitamin D and calcium in type 2 diabetes. A systematic review and meta-analysis. J Clin Endocrinol Metab. 2007 Jun;92(6):2017-29. doi: 10.1210/jc.2007-0298. Epub 2007 Mar 27. PMID 17389701
- [Background] Ford ES, Ajani UA, McGuire LC, Liu S. Concentrations of serum vitamin D and the metabolic syndrome among U.S. adults. Diabetes Care. 2005 May;28(5):1228-30. doi: 10.2337/diacare.28.5.1228. No abstract available. PMID 15855599
- [Background] Nagpal J, Pande JN, Bhartia A. A double-blind, randomized, placebo-controlled trial of the short-term effect of vitamin D3 supplementation on insulin sensitivity in apparently healthy, middle-aged, centrally obese men. Diabet Med. 2009 Jan;26(1):19-27. doi: 10.1111/j.1464-5491.2008.02636.x. PMID 19125756
- [Background] Fliser D, Stefanski A, Franek E, Fode P, Gudarzi A, Ritz E. No effect of calcitriol on insulin-mediated glucose uptake in healthy subjects. Eur J Clin Invest. 1997 Jul;27(7):629-33. doi: 10.1046/j.1365-2362.1997.1520699.x. PMID 9263752
- [Background] Pittas AG, Harris SS, Stark PC, Dawson-Hughes B. The effects of calcium and vitamin D supplementation on blood glucose and markers of inflammation in nondiabetic adults. Diabetes Care. 2007 Apr;30(4):980-6. doi: 10.2337/dc06-1994. Epub 2007 Feb 2. PMID 17277040
- [Background] Gannage-Yared MH, Azoury M, Mansour I, Baddoura R, Halaby G, Naaman R. Effects of a short-term calcium and vitamin D treatment on serum cytokines, bone markers, insulin and lipid concentrations in healthy post-menopausal women. J Endocrinol Invest. 2003 Aug;26(8):748-53. doi: 10.1007/BF03347358. PMID 14669830
- [Background] Fay TN, Jacobs I, Teisner B, Poulsen O, Chapman MG, Stabile I, Bohn H, Westergaard JG, Grudzinskas JG. Two fetal antigens (FA-1 and FA-2) and endometrial proteins (PP12 and PP14) isolated from amniotic fluid; preliminary observations in fetal and maternal tissues. Eur J Obstet Gynecol Reprod Biol. 1988 Sep;29(1):73-85. doi: 10.1016/0028-2243(88)90167-0. PMID 3224746
- [Background] Abdallah BM, Jensen CH, Gutierrez G, Leslie RG, Jensen TG, Kassem M. Regulation of human skeletal stem cells differentiation by Dlk1/Pref-1. J Bone Miner Res. 2004 May;19(5):841-52. doi: 10.1359/JBMR.040118. Epub 2004 Jan 19. PMID 15068508
- [Background] Abdallah BM, Boissy P, Tan Q, Dahlgaard J, Traustadottir GA, Kupisiewicz K, Laborda J, Delaisse JM, Kassem M. dlk1/FA1 regulates the function of human bone marrow mesenchymal stem cells by modulating gene expression of pro-inflammatory cytokines and immune response-related factors. J Biol Chem. 2007 Mar 9;282(10):7339-51. doi: 10.1074/jbc.M607530200. Epub 2006 Dec 19. PMID 17182623
- [Background] Snijder MB, van Dam RM, Visser M, Deeg DJ, Dekker JM, Bouter LM, Seidell JC, Lips P. Adiposity in relation to vitamin D status and parathyroid hormone levels: a population-based study in older men and women. J Clin Endocrinol Metab. 2005 Jul;90(7):4119-23. doi: 10.1210/jc.2005-0216. Epub 2005 Apr 26. PMID 15855256
- [Background] Vieth R. Vitamin D toxicity, policy, and science. J Bone Miner Res. 2007 Dec;22 Suppl 2:V64-8. doi: 10.1359/jbmr.07s221. PMID 18290725
- [Background] Maalouf J, Nabulsi M, Vieth R, Kimball S, El-Rassi R, Mahfoud Z, El-Hajj Fuleihan G. Short- and long-term safety of weekly high-dose vitamin D3 supplementation in school children. J Clin Endocrinol Metab. 2008 Jul;93(7):2693-701. doi: 10.1210/jc.2007-2530. Epub 2008 Apr 29. PMID 18445674
- [Background] Richter V, Rassoul F, Purschwitz K, Hentschel B, Reuter W, Kuntze T. Circulating vascular cell adhesion molecules VCAM-1, ICAM-1, and E-selectin in dependence on aging. Gerontology. 2003 Sep-Oct;49(5):293-300. doi: 10.1159/000071710. PMID 12920349
- [Background] Bluher M, Bullen JW Jr, Lee JH, Kralisch S, Fasshauer M, Kloting N, Niebauer J, Schon MR, Williams CJ, Mantzoros CS. Circulating adiponectin and expression of adiponectin receptors in human skeletal muscle: associations with metabolic parameters and insulin resistance and regulation by physical training. J Clin Endocrinol Metab. 2006 Jun;91(6):2310-6. doi: 10.1210/jc.2005-2556. Epub 2006 Mar 21. PMID 16551730
- [Derived] Bacha DS, Rahme M, Al-Shaar L, Baddoura R, Halaby G, Singh RJ, Mahfoud ZR, Habib R, Arabi A, El-Hajj Fuleihan G. Vitamin D3 Dose Requirement That Raises 25-Hydroxyvitamin D to Desirable Level in Overweight and Obese Elderly. J Clin Endocrinol Metab. 2021 Aug 18;106(9):e3644-e3654. doi: 10.1210/clinem/dgab296. PMID 33954783
- [Derived] El Sabeh M, Ghanem P, Al-Shaar L, Rahme M, Baddoura R, Halaby G, Singh RJ, Vanderschueren D, Bouillon R, El-Hajj Fuleihan G. Total, Bioavailable, and Free 25(OH)D Relationship with Indices of Bone Health in Elderly: A Randomized Controlled Trial. J Clin Endocrinol Metab. 2021 Jan 23;106(2):e990-e1001. doi: 10.1210/clinem/dgaa780. PMID 33280041
- [Derived] Bassatne A, Jafari A, Kassem M, Mantzoros C, Rahme M, El-Hajj Fuleihan G. Delta-like 1 (DLK1) is a possible mediator of vitamin D effects on bone and energy metabolism. Bone. 2020 Sep;138:115510. doi: 10.1016/j.bone.2020.115510. Epub 2020 Jul 1. PMID 32622071
- [Derived] Rahme M, Al-Shaar L, Singh R, Baddoura R, Halaby G, Arabi A, Habib RH, Daher R, Bassil D, El-Ferkh K, Hoteit M, El-Hajj Fuleihan G. Limitations of platform assays to measure serum 25OHD level impact on guidelines and practice decision making. Metabolism. 2018 Dec;89:1-7. doi: 10.1016/j.metabol.2018.09.003. Epub 2018 Sep 15. PMID 30227144
- [Derived] Arabi A, Khoueiry-Zgheib N, Awada Z, Mahfouz R, Al-Shaar L, Hoteit M, Rahme M, Baddoura R, Halabi G, Singh R, El Hajj Fuleihan G. CYP2R1 polymorphisms are important modulators of circulating 25-hydroxyvitamin D levels in elderly females with vitamin insufficiency, but not of the response to vitamin D supplementation. Osteoporos Int. 2017 Jan;28(1):279-290. doi: 10.1007/s00198-016-3713-5. Epub 2016 Jul 30. PMID 27473187
- [Derived] El-Hajj Fuleihan G, Baddoura R, Habib RH, Halaby G, Arabi A, Rahme M, Singh RJ, Kassem M, Mahfoud Z, Hoteit M, Daher RT, Kassir MF. Effect of vitamin D replacement on indexes of insulin resistance in overweight elderly individuals: a randomized controlled trial. Am J Clin Nutr. 2016 Aug;104(2):315-23. doi: 10.3945/ajcn.116.132589. Epub 2016 Jul 13. PMID 27413130